CLINICAL TRIAL: NCT01501552
Title: Randomised Controlled Trial Testing the Incremental Effect of Strategies That Raise Awareness, Acceptance and Performance of Identification and Brief Intervention Programmes for Harmful Alcohol Consumption in Primary Health Care
Brief Title: Trial Testing the Effect of Strategies on Performance of Brief Intervention Programmes for Harmful Alcohol Consumption
Acronym: ODHIN_RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: European Commission (Other); Stichting Katholieke Universiteit (Other); University of Newcastle Upon-Tyne (Other); King's College London (Other); Göteborg University (Other); Linkoeping University (Other Government); Department of Health, Generalitat de Catalunya (Other Government); State Agency for Solving Alcohol Problems (Other); University College, London (Other); Maastricht University (Other); Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Antoni Gual, Head of the Alcohol Unit, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: ECGA259268
Record Dates: First submitted 2011-12-16; First posted 2011-12-29 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Alcoholism
Keywords: Primary health care; Identification and Brief Intervention Programmes; Hazardous and harmful alcohol consumption
MeSH Terms: conditions — Alcoholism | interventions — Palliative Care; Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Treatment as usual (No Intervention): In the no-intervention treatment as usual group, a package, containing a summary card of the national guideline recommendation, will be delivered to each provider unit without demonstration. In Poland, the summary card will be adapted from the PHEPA guidelines (ref) for the purposes of this trial. The treatment as usual group will be requested to screen and offer person-to-person SBI at the PHCU.
- Training & support (T&S) (Experimental): The T&S only group will be offered two face-to-face educational meetings of at least one hour and a maximum of 2 hours, and one telephone support call of at least ten minutes and a maximum of 30 minutes. The telephone call will be offered to one of the GPs ('leader'). Depending on the needs of the PHCU, one additional face to face training (1 to 2 hours) may be offered. The time interval between meetings will be on average 2 weeks. The training sessions will address improving knowledge, skills, attitudes, and perceived barriers and facilitators by combining theory and practice-based training.
  Interventions: Other: Training and support (T&S)
- Financial incentive (Experimental): The financial incentive only group will receive a financial incentive depending on their screening and brief intervention activities. They will be paid for the performance, with the country dependent system of pay (fee for item or fee for achieving set rates) and based on normal practices and financial rates for financial incentives for clinical preventive activities.
  Interventions: Other: Financial incentive
- E-SBI (Experimental): The e-SBI (online screening and brief intervention)only group are expected to refer identified at-risk patients to an approved e-SBI programme, which will be either country specific (where these exist) or based on the WHO e-SBI programme (Poland).
  Interventions: Other: E-SBI (online screening and brief intervention)
- T&S and financial incentive (Experimental): The T&S and financial incentive group will be offered two face-to-face educational meetings of at least one hour and a maximum of 2 hours, and one telephone support call of at least ten minutes and a maximum of 30 minutes. Also, they will receive a financial incentive depending on their screening and brief intervention activities. They will be paid for the performance, with the country dependent system of pay (fee for item or fee for achieving set rates) and based on normal practices and financial rates for financial incentives for clinical preventive activities.
  Interventions: Other: Training and support (T&S); Other: Financial incentive
- T&S and e-SBI (Experimental): The T&S and e-SBI group will be offered two face-to-face educational meetings of at least one hour and a maximum of 2 hours, and one telephone support call of at least ten minutes and a maximum of 30 minutes. The telephone call was offered to one of the GPs ('leader'). Depending on the needs of the PHCU, one additional face to face training (1 to 2 hours) was offered. Also this group is expected to refer identified at-risk patients to an approved e-SBI (online screening and brief intervention) programme, which will either be country specific (where these exist) or based on the WHO e-SBI programme (Poland).
  Interventions: Other: Training and support (T&S); Other: E-SBI (online screening and brief intervention)
- Financial incentive and e-SBI (Experimental): The financial incentive and e-SBI (online screening and brief intervention) group will be paid for screening and referral performance instead of actual delivery of e-SBI by themselves as in line with the e-SBI only group, with the country dependent system of pay (fee for item or fee for achieving set rates) and based on normal practices and financial rates for financial incentives for clinical preventive activities.
  Interventions: Other: Financial incentive; Other: E-SBI (online screening and brief intervention)
- T&S, financial incentive and e-SBI (Experimental): The T&S, financial incentive and e-SBI (online screening and brief intervention) group will be offered two face-to-face educational meetings of at least one hour and a maximum of 2 hours, and one telephone support call of at least ten minutes and a maximum of 30 minutes. The telephone call will be offered to one of the GPs ('leader'). Also, they are expected to offer screening at the PHCU and to refer screen positive patients to e-SBI programmes. Additionally, they will be paid for screening and referral performance, with the country dependent system of pay (fee for item or fee for achieving set rates) and based on normal practices and financial rates for financial incentives for clinical preventive activities.
  Interventions: Other: Training and support (T&S); Other: Financial incentive; Other: E-SBI (online screening and brief intervention)

INTERVENTIONS:
Other: Training and support (T&S) — Two face-to-face educational meetings of at least one hour and a maximum of 2 hours, and one telephone support call of at least ten minutes and a maximum of 30 minutes. The telephone call will be offered to one of the GPs ('leader'). Depending on the needs of the PHCU, one additional face to face training (1 to 2 hours) may be offered. The time interval between meetings will be on average 2 weeks. The training sessions will address improving knowledge, skills, attitudes, and perceived barriers and facilitators by combining theory and practice-based training.
  Arms: T&S and e-SBI; T&S and financial incentive; T&S, financial incentive and e-SBI; Training & support (T&S)
Other: Financial incentive — Groups will receive a financial incentive depending on their screening and brief intervention activities. They will be paid for the performance, with the country dependent system of pay (fee for item or fee for achieving set rates) and based on normal practices and financial rates for financial incentives for clinical preventive activities.
  Arms: Financial incentive; Financial incentive and e-SBI; T&S and financial incentive; T&S, financial incentive and e-SBI
Other: E-SBI (online screening and brief intervention) — Referring identified at-risk patients to an approved e-SBI programme, which will be either country specific (where these exist) or based on the WHO e-SBI programme (Poland).
  Arms: E-SBI; Financial incentive and e-SBI; T&S and e-SBI; T&S, financial incentive and e-SBI

SUMMARY:
The overall objective is to study if training and support, financial reimbursement and referral to an internet based brief intervention programme, singly or in combination, may increase implementation of evidence based methods of identification and brief intervention for excessive alcohol consumption in routine primary health care.

DETAILED DESCRIPTION:
The study will be a stepped cluster RCT in 5 countries and the endpoint of the study is the number of interventions delivered during a certain time period. More specifically, the RCT will examine:

* The effect of Continuous Medical Education (CME) to PHC providers
* The effect of financial reimbursement to PHC providers as a pay-for-performance of brief alcohol interventions
* Whether an alternative internet based method of delivering brief intervention can increase the proportion of patients reached
* If one implementation strategy will give an added value to one already enforced.

ELIGIBILITY:
Inclusion Criteria:

* Primary Health Care Units (PHCU) of approximate size of 5.000-20.000 registered patients
* Primary Health Care Units (PHCU) located in Spain, Poland, Sweden, England or The Netherlands
* Providers must be physicians or nurses

Exclusion Criteria:

* Primary Health Care Units with less than 5.000 registered patients or over 20.000 registered patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of screening tests carried out in primary health care settings to detect excessive alcohol consumption care | 5 months
  Screening rates will be calculated at five time points: during a four week period during the third month before the start of the study (baseline measurement), in three consecutive four week blocks during the twelve week intervention period (intervention measurement) and during a four week block during the sixth month after the end of the intervention period (follow-up measurement).
Number of brief interventions for excessive alcohol consumption delivered in primary health care settings | 5 months
  Brief intervention rates will be calculated at five time points: during a four week period during the third month before the start of the study (baseline measurement), in three consecutive four week blocks during the twelve week intervention period (intervention measurement) and during a four week block during the sixth month after the end of the intervention period (follow-up measurement).

SECONDARY OUTCOMES:
Level of role security of primary health care providers measured by their answers to the SAAPPQ instrument | 3 months
  Role security of the primary health care providers will be measured through their responses to the SAAPPQ (a validated instrument based on factor analysis (Anderson & Clement 1987) of the original alcohol and alcohol problems perception questionnaire developed and validated by Cartwright (1980))at three time points: baseline, end of intervention period, and follow-up.
Level of therapeutic commitment of primary health care providers measured by their answers to the SAAPPQ instrument | 3 months
  Therapeutic commitment of the primary health care providers will be measured through their responses to the SAAPPQ (a validated instrument based on factor analysis (Anderson & Clement 1987) of the original alcohol and alcohol problems perception questionnaire developed and validated by Cartwright (1980))at three time points: baseline, end of intervention period, and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Preben - Bendtsen, MD, Principal Investigator — Linkoeping University; Fredrik - Spak, MD, Principal Investigator — Göteborg University; Peter - Anderson, MD, Principal Investigator — Maastricht University
Locations (10):
- Netherlands (2):
  - Maastricht University, Maastricht, Netherlands
  - Stichting Katholieke Universiteit, Nijmegen, Netherlands
- Poland (2):
  - Pomorski Uniwersytet Medyczny w Szczecinie, Szczecin, Poland
  - Panstwowa Agencja Rozwiazywania Problemow Alkoholowych, Warsaw, Poland
- Departament de Salut de la Generalitat de Catalunya, Barcelona, Catalonia, Spain
- Sweden (2):
  - Goeteborgs Universitet, Gothenburg, Sweden
  - Linköping University, Linköping, Sweden
- United Kingdom (3):
  - King's College London, London, England
  - University College, London, London, England
  - University of Newcastle Upon-Tyne, Newcastle upon Tyne, England

REFERENCES:
- [Derived] Angus C, Li J, Romero-Rodriguez E, Anderson P, Parrott S, Brennan A. Cost-effectiveness of strategies to improve delivery of brief interventions for heavy drinking in primary care: results from the ODHIN trial. Eur J Public Health. 2019 Apr 1;29(2):219-225. doi: 10.1093/eurpub/cky181. PMID 30239676
- [Derived] Anderson P, Kloda K, Kaner E, Reynolds J, Bendtsen P, Pelgrum-Keurhorst MN, Segura L, Wojnar M, Mierzecki A, Deluca P, Newbury-Birch D, Parkinson K, Okulicz-Kozaryn K, Drummond C, Laurant MGH, Gual A. Impact of practice, provider and patient characteristics on delivering screening and brief advice for heavy drinking in primary healthcare: Secondary analyses of data from the ODHIN five-country cluster randomized factorial trial. Eur J Gen Pract. 2017 Dec;23(1):241-245. doi: 10.1080/13814788.2017.1374365. PMID 29022763
- [Derived] Anderson P, Coulton S, Kaner E, Bendtsen P, Kloda K, Reynolds J, Segura L, Wojnar M, Mierzecki A, Deluca P, Newbury-Birch D, Parkinson K, Okulicz-Kozaryn K, Drummond C, Gual A. Delivery of Brief Interventions for Heavy Drinking in Primary Care: Outcomes of the ODHIN 5-Country Cluster Randomized Trial. Ann Fam Med. 2017 Jul;15(4):335-340. doi: 10.1370/afm.2051. PMID 28694269
- [Derived] Keurhorst M, Anderson P, Heinen M, Bendtsen P, Baena B, Brzozka K, Colom J, Deluca P, Drummond C, Kaner E, Kloda K, Mierzecki A, Newbury-Birch D, Okulicz-Kozaryn K, Palacio-Vieira J, Parkinson K, Reynolds J, Ronda G, Segura L, Slodownik L, Spak F, van Steenkiste B, Wallace P, Wolstenholme A, Wojnar M, Gual A, Laurant M, Wensing M. Impact of primary healthcare providers' initial role security and therapeutic commitment on implementing brief interventions in managing risky alcohol consumption: a cluster randomised factorial trial. Implement Sci. 2016 Jul 16;11:96. doi: 10.1186/s13012-016-0468-5. PMID 27422283
- [Derived] Bendtsen P, Mussener U, Karlsson N, Lopez-Pelayo H, Palacio-Vieira J, Colom J, Gual A, Reynolds J, Wallace P, Segura L, Anderson P. Implementing referral to an electronic alcohol brief advice website in primary healthcare: results from the ODHIN implementation trial. BMJ Open. 2016 Jun 16;6(6):e010271. doi: 10.1136/bmjopen-2015-010271. PMID 27311902
- [Derived] Keurhorst M, Heinen M, Colom J, Linderoth C, Mussener U, Okulicz-Kozaryn K, Palacio-Vieira J, Segura L, Silfversparre F, Slodownik L, Sorribes E, Laurant M, Wensing M. Strategies in primary healthcare to implement early identification of risky alcohol consumption: why do they work or not? A qualitative evaluation of the ODHIN study. BMC Fam Pract. 2016 Jun 7;17:70. doi: 10.1186/s12875-016-0461-8. PMID 27267887
- [Derived] Anderson P, Bendtsen P, Spak F, Reynolds J, Drummond C, Segura L, Keurhorst MN, Palacio-Vieira J, Wojnar M, Parkinson K, Colom J, Kloda K, Deluca P, Baena B, Newbury-Birch D, Wallace P, Heinen M, Wolstenholme A, van Steenkiste B, Mierzecki A, Okulicz-Kozaryn K, Ronda G, Kaner E, Laurant MG, Coulton S, Gual T. Improving the delivery of brief interventions for heavy drinking in primary health care: outcome results of the Optimizing Delivery of Health Care Intervention (ODHIN) five-country cluster randomized factorial trial. Addiction. 2016 Nov;111(11):1935-1945. doi: 10.1111/add.13476. Epub 2016 Jul 25. PMID 27237081
- [Derived] Keurhorst MN, Anderson P, Spak F, Bendtsen P, Segura L, Colom J, Reynolds J, Drummond C, Deluca P, van Steenkiste B, Mierzecki A, Kloda K, Wallace P, Newbury-Birch D, Kaner E, Gual T, Laurant MG. Implementing training and support, financial reimbursement, and referral to an internet-based brief advice program to improve the early identification of hazardous and harmful alcohol consumption in primary care (ODHIN): study protocol for a cluster randomized factorial trial. Implement Sci. 2013 Jan 24;8:11. doi: 10.1186/1748-5908-8-11. PMID 23347874
- See also: Optimizing delivery of health interventions project's website. — http://www.odhinproject.eu